CLINICAL TRIAL: NCT05714267
Title: The Effect of Noise Control and Music Therapy on Anxiety, Vital Signs and Post-Operative Pain in Total Knee Prosthesis Surgery
Brief Title: Effect of Noise Control During Total Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: Bvu_Nursing-1
Record Dates: First submitted 2021-07-05; First posted 2023-02-06 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Knee Osteoarthritis
Keywords: Music therapy; Active noise control; Pasive noise control; Knee replacement
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Music Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Active noise cancelling (Experimental): Patients corresponding to the number 1 blocks in the randomization table according to the order of surgery were included in the active noise control group. Preoperative care of the patients was performed by clinical nurses. After transferring to the operating room and performing spinal anesthesia, the active noise control headset (Sony WH1000xm4) was placed on the patient's head. The active noise control feature of the headset was turned on and it was not removed until the dressing of the patient was closed at the end of the operation. In this group, the vital signs of the patients were followed up during the surgery. At the end of each surgery, the researcher disinfected the earplugs with an antiseptic solution containing 2% chlorhexidine. In addition, the battery level of the headset was checked and charged by the researcher when necessary. This ensures that the headset is ready for the next patient.
  Interventions: Device: Active noise cancelling
- Passive noise cancelling (Experimental): The patients corresponding to the number 2 blocks in the randomization table according to the order of operation were included in the passive noise control group. Preoperative care of the patients was performed by clinical nurses. After transferring to the operating room and performing spinal anesthesia, passive noise control headset (3M Peltor Optime II) was placed on the patient's head. The earphone was not removed until the dressing of the patient was closed at the end of the surgery. In this group, the vital signs of the patients were followed up during the surgery. At the end of each operation, the earplugs were disinfected by the researcher with an antiseptic solution containing 2% chlorhexidine and prepared for the next patient.
  Interventions: Device: Passive noice cancelling
- Active noise cancelling with music therapy (Experimental): Patients corresponding to blocks numbered 3 in the randomization table according to the order of surgery were included in the music therapy group. Preoperative care of the patients was performed by clinical nurses. After transferring to the operating room and performing spinal anesthesia, the headset (Sony WH1000xm4) was positioned on the patient's head as shown in Figure 3.7-5 (A). iPod Touch 7th Generation music player with Spotify mobile application was used for music application. The connection between the headset and the music player was provided via Bluetooth. Music chosen by the patient; Active noise control was turned on and the patient was listened to until the dressing was removed at the end of the operation. The vital signs of the patient during the operation were followed up. In addition, the battery level of the headset was checked and charged by the researcher when necessary. This ensures that the headset is ready for the next patient.
  Interventions: Device: Active noise cancelling with music therapy
- Control group (No Intervention): Patients corresponding to blocks numbered 0 in the randomization table according to the order of surgery were included in the control group. The patients, whose preoperative care was performed by clinical nurses, were transferred to the operating room and spinal anesthesia was administered. No intervention was made in this group during the surgery. The vital signs of the patients were followed up during the operation.

INTERVENTIONS:
Device: Active noise cancelling — During the operation, active noise canceling device (Sony wh100xm3) will be applied to the patients in Group-1 after spinal anesthesia is applied and will not be removed until the operation is completed. At the end of the surgery, the trait anxiety scale will be administered to the patients and the VAS pain scale will be administered at the 1st Hour, 8th Hour and 24th Hour. The obtained data will be recorded.
  Arms: Active noise cancelling
Device: Passive noice cancelling — During the operation, passive noise canceling device (3M Peltor X5a) will be applied to the patients in Group-2 after spinal anesthesia is applied and will not be removed until the operation is completed. At the end of the surgery, the trait anxiety scale will be administered to the patients and the VAS pain scale will be administered at the 1st Hour, 8th Hour and 24th Hour. The obtained data will be recorded.
  Arms: Passive noise cancelling
Device: Active noise cancelling with music therapy — The patients in Group-3 will be given music therapy with an active noise canceling tool (Sony wh100xm3) during the surgery. The music that the patient will listen to will be left to the patient's preference. Music therapy with an active noise canceling device will be applied after spinal anesthesia is applied and will not be removed until the surgery is completed. At the end of the surgery, the trait anxiety scale will be administered to the patients and the VAS pain scale will be administered at the 1st Hour, 8th Hour and 24th Hour. The obtained data will be recorded.
  Arms: Active noise cancelling with music therapy

SUMMARY:
Music has emerged as a well-received medical intervention. Patients may be uncomfortable during total joint replacement, which can result in high sedation requirements. These requirements put patients at risk of surgical stress. This study compares the effect of passive noise-cancellation versus active noise cancellation with music on pain, vital signs and anxiety during elective total knee replacement.

DETAILED DESCRIPTION:
Unwanted sound that mixes with the sounds being listened to is defined as noise, and the sound community formed by the combination of many noise sources is defined as noise pollution. Environmental noise has many negative effects on human health, such as increasing stress and anxiety, causing the development of cerebral and cardiovascular diseases, and creating a risk of hearing loss.

Today, it is reported that noise pollution in hospitals has increased exponentially compared to previous years . It is reported that the noise is especially at high levels in the operating room units of hospitals and frequently exceeds both the 30 dBA (Decibel A) threshold determined by the World Health Organization and the American Occupational Safety and Health Administration standard. When we look at the studies in which the environmental noise in the operating room environment is examined, it is seen that the noise level varies between 80 and 119 dBA. These noise ranges are determined for both patient and employee health. is beyond the limits.

The noise that patients are exposed to in operating rooms can be caused by both healthcare workers and operating room equipment. Perioperative Nurses Association (AORN) created the "AORN Guide on Managing Distraction and Noise During Perioperative Patient Care" in 2014 to draw attention to the problem of loud noise in the operating room. According to this guideline, updated in 2020, noise is a risky situation that interrupts intraoperative care. For this reason, it is reported that noise should be prevented with an inter-team approach in order for effective care and treatment to continue. In the AORN report, it is reported that among the sources of noise are monitors, ventilators, air conditioning systems, telephones, pagers, surgical equipment, anesthesia devices, conversations within the team, and loud music. The methods used in surgeries and the choice of surgical instruments also affect noise levels. For this reason, it can be said that noise levels may change in surgeries performed with different instruments in different parts of the body. Especially in knee and hip replacement surgeries, when tools such as oscillator saws, hammers and surgical drills, which are used to shape the joint and replace the joint prosthesis, are used during the operation, it creates a higher noise compared to other surgeries. Simpson reported in their study that the noise level of the instruments used during knee and hip replacement surgery increased up to 105 decibels. While this noise level is equivalent to the noise heard while waiting next to a working helicopter, it is well above the thresholds recommended by NIOSH, OSHA and WHO.

It is reported that the negative effects of environmental noise during surgery on patients are controlled with sedative agents given to the patient during surgery. In addition, it is known that patients are made to listen to music to reduce the effect of environmental noise and to relax the patient. When the studies are examined, it is seen that there are limitations in both methods used. Listening to louder music so that the high-frequency sounds that occur during prosthetic surgeries are not heard by the patients can be another source of anxiety for the patients. Sedative opioid agents given to calm patients pose various risks, such as respiratory depression, death or permanent brain damage, and this is defined as a patient safety problem in the literature. Since the degeneration (arthrosis) of the knee joint will occur over the years, the patient population in need of prosthesis is generally geriatric. This situation causes the adverse risks of sedation on elderly patients to be much higher. The operating room nurse should take the necessary measures to reduce the stress, fear and anxiety of the patient who will undergo surgery. It is one of the independent roles of the nurse to ensure that non-pharmacological methods are used instead of pharmacological sedative agents applied to the patient.

Active noise control is one of the methods in which the noise is controlled with headphones that produce a sound in phase opposite to the environmental noise, and passive noise control is one of the methods in which the noise is controlled by the isolation method. Music therapy, on the other hand, lowers the blood pressure and pulse of the patients, regulates the respiratory rate and increases the oxygen saturation.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18-80
* To participate in the research voluntarily,
* To be able to read and write Turkish,
* American Association of Anesthesiologists (ASA) classification I or II,
* To have total knee arthroplasty surgery due to joint degeneration (gonarthrosis),
* Not using any medication that will affect anxiety,
* To be problem-free in terms of sensory perceptions and communication,
* The patient is conscious, oriented and cooperative.

Exclusion Criteria:

* Having a total knee replacement surgery due to an acquired physical trauma to the knee joint,
* Presence of diagnosed cancer in the patient.
* Being diagnosed with any psychiatric illness,
* Having previously undergone arthroplasty surgery (Revision arthroplasty).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-08-04 (Actual)

PRIMARY OUTCOMES:
State and trait anxiety scale | Before the surgery
  The application period of the scale, which can be applied to all individuals over the age of 14, is ten minutes on average. With the State Anxiety Scale, the individual can evaluate his feelings in a certain place and time according to 20 statements. By using the trait anxiety scale, the feelings of the individual can be evaluated according to these 20 expressions, regardless of the circumstances. The total weighted score for the reverse statements is subtracted from the total weight score for direct statements, and a constant value is added to this number. This value is 50 for the state anxiety scale and 35 for the trait anxiety scale. Both scales are scored between 20-80. A high score indicates high anxiety.
Visual Analog Scale | Change from baseline to 1 months
  Visual Analogue Scale (VAS) was used to evaluate the assumed pain differences between groups. In order to measure the severity of pain with VAS, a 10 cm long ruler was used, in the range of 0-10 points, with "No pain" on one end and "Unbearable pain" on the other end. The patient was told that he was free to mark any part of the ruler, including 0-10. Then, the patient was asked to mark a point showing the severity of the pain on the created ruler. Numerical data were obtained by measuring in centimeters between the zero point of the ruler and the point marked by the patient. The numerical value corresponding to the point marked by the patient on the VAS was recorded in the data collection form. patient's pain;
  1. Before surgery,
  2. Immediately after the operation,
  3. 8 hours after surgery
  4. It was evaluated 4 times, 24 hours after the surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Deniz Öztekin, Professor, Study Director — Doğuş University
Locations (1):
- Bezmialem University, Istanbul, Fatih, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Basner M, Babisch W, Davis A, Brink M, Clark C, Janssen S, Stansfeld S. Auditory and non-auditory effects of noise on health. Lancet. 2014 Apr 12;383(9925):1325-1332. doi: 10.1016/S0140-6736(13)61613-X. Epub 2013 Oct 30. PMID 24183105
- [Background] Tran BW, Nowrouz MY, Dhillon SK, Xie KK, Breslin KM, Golladay GJ. The Impact of Music and Noise-Cancellation on Sedation Requirements During Total Knee Replacement: A Randomized Controlled Trial. Geriatr Orthop Surg Rehabil. 2020 Mar 4;11:2151459320910844. doi: 10.1177/2151459320910844. eCollection 2020. PMID 32181048
- [Background] Liu M, Yi C, Yin F, Dai Y. Noise in the outpatient operating room. Gland Surg. 2020 Apr;9(2):380-384. doi: 10.21037/gs.2020.04.09. PMID 32420262
- [Background] Yeganeh S, Torabizadeh C, Bahmani T, Molazem Z, Doust HY, Dehnavi SD. Examining the views of operating room nurses and physicians on the relationship between professional values and professional communication. BMC Nurs. 2022 Jan 14;21(1):17. doi: 10.1186/s12912-021-00778-x. PMID 35031042
- [Background] Wang X, Zeng L, Li G, Xu M, Wei B, Li Y, Li N, Tao L, Zhang H, Guo X, Zhao Y. A cross-sectional study in a tertiary care hospital in China: noise or silence in the operating room. BMJ Open. 2017 Sep 18;7(9):e016316. doi: 10.1136/bmjopen-2017-016316. PMID 28928180
- [Background] Sampieri G, Namavarian A, Levin M, Philteos J, Lee JW, Koskinen A, Lin V, Lee J. Noise in Otolaryngology - Head and Neck Surgery operating rooms: a systematic review. J Otolaryngol Head Neck Surg. 2021 Feb 11;50(1):8. doi: 10.1186/s40463-020-00487-6. PMID 33573705
- [Background] Martinez-Millana A, Lizondo A, Gatta R, Vera S, Salcedo VT, Fernandez-Llatas C. Process Mining Dashboard in Operating Rooms: Analysis of Staff Expectations with Analytic Hierarchy Process. Int J Environ Res Public Health. 2019 Jan 11;16(2):199. doi: 10.3390/ijerph16020199. PMID 30642000
- [Background] Grozdanovic D, Janackovic GL, Grozdanovic M, Mitkovic MB, Mitkovic MM. The Selection of Main Surgical Work Factors in Operating Rooms. Inquiry. 2021 Jan-Dec;58:469580211067497. doi: 10.1177/00469580211067497. PMID 34908506
- [Background] Song JJ, Vanneste S, De Ridder D. Dysfunctional noise cancelling of the rostral anterior cingulate cortex in tinnitus patients. PLoS One. 2015 Apr 13;10(4):e0123538. doi: 10.1371/journal.pone.0123538. eCollection 2015. PMID 25875099
- [Background] Zangari S, Mirowsky JE. A simple, cost-effective, and novel method for determining the efficiency of industrial and commercial noise-canceling earmuffs. Noise Health. 2019 May-Jun;21(100):108-115. doi: 10.4103/nah.NAH_52_19. PMID 32655064
- [Background] Ghaleb FA, Kamat MB, Salleh M, Rohani MF, Abd Razak S. Two-stage motion artefact reduction algorithm for electrocardiogram using weighted adaptive noise cancelling and recursive Hampel filter. PLoS One. 2018 Nov 20;13(11):e0207176. doi: 10.1371/journal.pone.0207176. eCollection 2018. PMID 30457996
- See also: Asco Battery Operated Cannulated Drill Machine, For Industrial — https://www.indiamart.com/proddetail/battery-operated-cannulated-drill-machine-4420781412.html.
- See also: Orthopedic Mallet — https://bossinstruments.com/product/7-orthopedic-mallet-2lb-solid-head/